CLINICAL TRIAL: NCT01546753
Title: Walnut Oral Immunotherapy for Tree Nut Allergy
Acronym: WOIT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113364; FARE (Other: Food Allergy Research and Education)
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: Tree Nut Allergy
Keywords: Walnut allergy; Tree nut allergy; Oral immunotherapy; Food allergy; Desensitization; Sustained unresponsiveness
MeSH Terms: conditions — Nut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 2:1 ratio to either active treatment (final dose 1500mg walnut protein (WP), n=20) or placebo (n=10). Subjects will do a 1-day desensitization to enable subjects to tolerate 6 mg of WP or placebo (initial day escalation). After the initial escalation day obtaining at least 1.5mg and up to 6mg of WP or placebo, dosing build-up will be every 2 wks thru dose 24 (34 wks). A maintenance dose will be given for 4 wks, then a 5g protein OFC to walnut & a 5g protein OFC to a 2nd tree nut (~38 wks), then the study will be unblinded. Placebo subjects that fail the OFC will cross-over to active treatment and escalate to 1500mg target dose. Subjects will be followed for 298 wks (~6 yrs) total on active treatment including an OFC (both on & off therapy) to walnut and 2nd tree nut at 142 wk & end of study. Subjects with reduced serum specific IgE to <5kU/L to walnut and 2nd tree nut at yearly visits before the end of study at 298 wks are eligible for a tolerance OFC.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Walnut Protein Powder (Experimental): 38 weeks on active walnut powder on blinded treatment phase
  Interventions: Drug: Walnut Protein Powder
- Oat Powder (Placebo Comparator): 38 weeks on placebo (oat) powder during blinded treatment phase
  Interventions: Drug: Oat Powder (placebo)
- Open-label Walnut Protein Powder (Other): Open-label treatment with walnut protein powder up to week 298 of total treatment
  Interventions: Drug: Open-label Walnut Protein Powder

INTERVENTIONS:
Drug: Walnut Protein Powder — Blinded study product dosing begins with a 1-day oral desensitization protocol to walnut for subjects in the active arm. Starting at 0.1 mg protein and increasing to a maximum of 6 mg or until allergic symptoms develop. Subjects continue daily dosing of blinded OIT (walnut) with build-up every 2 weeks to a maximum daily dose of 1500mg at week 34, followed by 4 weeks of daily maintenance dosing. OFC to walnut and second tree nut occurs at week 38 then treatment is unblinded and open-label maintenance dosing occurs.
  Other Names: WOIT
  Arms: Walnut Protein Powder
Drug: Oat Powder (placebo) — Blinded study product dosing begins with a one-day oral desensitization protocol with placebo (oat) powder. Subjects in the placebo group will undergo the same protocol as those in the active group with placebo OIT dosing. Unblinding to treatment assignment will occur after the 38 week oral food challenge. Placebo subjects will cross-over to active, open-label treatment with walnut powder after the 38 week oral food challenge. beginning with initial escalation day, through build-up and maintenance dosing per the same protocol sequence as noted for active, walnut powder. Subjects will complete an oral food challenge to walnut and the second tree nut at week 38 then will continue on long-term, open-label maintenance dosing until the end of study using same protocol design.
  Other Names: Oat flour
  Arms: Oat Powder
Drug: Open-label Walnut Protein Powder — Open-label treatment phase begins after the 38 week oral food challenge with unblinding of treatment assignment. For those on active treatment, daily maintenance dosing occurs for up to a total of 298 weeks. For those on placebo treatment, cross-over to active, open-label treatment occurs using the same active treatment protocol. Placebo-crossover subjects will complete an oral food challenge to walnut and the second tree nut at week 38 of active therapy then continue on long-term, open-label maintenance dosing until the end of study using same protocol design. All subjects may reach a qualifying IgE to walnut/second tree nut early and will undergo an OFCs on and 4 weeks off OIT. All subjects will have OFCs on and 4 weeks off OIT at week 142 and at week 298, unless both walnut/second tree nut OFCs are passed at previous OFC prompting addition of these foods into the diet.
  Other Names: Open-label treatment
  Arms: Open-label Walnut Protein Powder

SUMMARY:
The purpose of this study is to determine if walnut oral immunotherapy can be used in participants allergic to tree nuts to reduce tree nut allergy and induce changes in the participant's immune system.

DETAILED DESCRIPTION:
Randomized, placebo controlled, Phase 1-2 study conducted at Arkansas Children's Hospital Research Institute (ACHRI) in tree nut allergic participants, ages 6-45 years with randomization following a 2:1 (active:placebo) format. The overall objectives were to evaluate the efficacy of walnut oral immunotherapy (WOIT) for induction of desensitization to walnut (secondary outcome) and a test tree nut (primary outcome) when compared to placebo after 38 weeks of treatment as assessed by double-blind, placebo-controlled food challenges (DBPCFC) to walnut and a test tree nut in tree nut allergic participants (defined by allergic reaction to </= 2 grams of walnut and test tree nut proteins during DBPCFC at study entry). Placebo participants were crossed-over to active therapy after unblinding at week 38. Participants were followed long-term (up to 6 years) on open-label WOIT treatment and assessed at yearly intervals based on pre-specified criteria for clinical outcomes of desensitization to walnut and a test tree nut (defined as safely consuming 5 grams of walnut and test tree nut protein during DBPCFC while on daily WOIT) and sustained unresponsiveness to walnut and a test tree nut (defined as safely consuming 5 grams of walnut and test tree nut protein during DBPCFC and 10 grams during an open feeding while off therapy for 4-6 weeks). Secondary outcomes were evaluated including safety and immune mechanistic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 45 years, either sex, any race, any ethnicity with a convincing clinical history of walnut or another tree nut allergy and either a positive prick skin test (≥ 3mm) or serologic evidence of allergic sensitization (defined as specific IgE > 0.35 kU/L) to walnut and at least one other tree nut.
* A positive 2000 mg oral food challenge at enrollment to walnut and to one other tree nut.
* Written informed consent from participant and/or parent/guardian
* Written assent from all subjects as appropriate
* All females of child bearing age must be using appropriate birth control

Exclusion Criteria:

* History of severe anaphylaxis to walnut or other tree nuts, defined as symptoms associated with hypoxia, hypotension or neurologic compromise (cyanosis or SpO2 < 92% at any stage, hypotension, confusion, collapse, loss of consciousness; or incontinence).
* Known allergy to oat
* Chronic disease (other than asthma, atopic dermatitis, rhinitis) requiring therapy or other respiratory or medical conditions deemed by the investigator to put the subject at increased risk of anaphylaxis or poor outcomes from receiving OIT or undergoing food challenge.
* Poor control or persistent activation of atopic dermatitis
* Active eosinophilic or other inflammatory (e.g., celiac) gastrointestinal disease in the past 2 years.
* Participation in any interventional study for food allergy in the past 6 months
* Participant is on "build-up phase" of immunotherapy (i.e., has not reached maintenance dosing).
* Severe asthma (2007 NHLBI Criteria Steps 5 or 6, see Appendix 2) or poorly controlled mild or moderate asthma
* Inability to discontinue antihistamines for initial day escalation, skin testing or OFC
* Use of omalizumab or other non-traditional forms of allergen immunotherapy (e.g., oral or sublingual) or immunomodulator therapy (not including corticosteroids) or biologic therapy within the past year
* Use of beta-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB) or calcium channel blockers
* Pregnancy or lactation

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2012-04-27 (Actual); Primary Completion 2015-07-02 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacie M Jones, MD, Principal Investigator — University of Arkansas for Medical Sciences / Arkansas Children's Hospital
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Jones SM, Pons L, Roberts JL, Scurlock AM, Perry TT, Kulis M, Shreffler WG, Steele P, Henry KA, Adair M, Francis JM, Durham S, Vickery BP, Zhong X, Burks AW. Clinical efficacy and immune regulation with peanut oral immunotherapy. J Allergy Clin Immunol. 2009 Aug;124(2):292-300, 300.e1-97. doi: 10.1016/j.jaci.2009.05.022. Epub 2009 Jul 3. PMID 19577283
- [Background] Hofmann AM, Scurlock AM, Jones SM, Palmer KP, Lokhnygina Y, Steele PH, Kamilaris J, Burks AW. Safety of a peanut oral immunotherapy protocol in children with peanut allergy. J Allergy Clin Immunol. 2009 Aug;124(2):286-91, 291.e1-6. doi: 10.1016/j.jaci.2009.03.045. Epub 2009 May 27. PMID 19477496
- [Background] Kulis M, Li Y, Lane H, Pons L, Burks W. Single-tree nut immunotherapy attenuates allergic reactions in mice with hypersensitivity to multiple tree nuts. J Allergy Clin Immunol. 2011 Jan;127(1):81-8. doi: 10.1016/j.jaci.2010.09.014. Epub 2010 Nov 18. PMID 21093029
- [Background] Varshney P, Jones SM, Scurlock AM, Perry TT, Kemper A, Steele P, Hiegel A, Kamilaris J, Carlisle S, Yue X, Kulis M, Pons L, Vickery B, Burks AW. A randomized controlled study of peanut oral immunotherapy: clinical desensitization and modulation of the allergic response. J Allergy Clin Immunol. 2011 Mar;127(3):654-60. doi: 10.1016/j.jaci.2010.12.1111. PMID 21377034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from allergy clinics, research databases and advertisement. Study recruitment occurred from April 2012 through September 2014.
Pre-assignment Details: Following consent and enrollment, screening included allergen skin testing, allergen-IgE testing, immune studies and DBPCFCs to placebo, walnut and at least one tree nut. Those meeting inclusion criteria were randomized 2:1 to blinded OIT (walnut vs. placebo) through week 38 when DBPCFCs were conducted. Unblinding of treatment assignment occurred at week 38; placebo subjects crossed over to active (walnut) OIT. OIT after week 38 was given daily as open-label treatment.
Groups:
- Walnut Protein Powder: Up to 298 weeks for active treatment subjects
  Walnut Protein Powder: Subjects randomized to the active treatment group begins with blinded study product (walnut) dosing utilizing a one-day oral desensitization protocol. Starting at 0.1 mg protein and increasing every thirty minutes until a maximum dose of 6 mg is reached or until allergic symptoms develop. After the initial escalation day, subjects will continue daily dosing with dosing build-every two weeks to a maximum dose of 1500mg walnut protein at 34 weeks. A daily maintenance dose (1500mg or the highest dose reached by 34 weeks) will be given for 4 weeks followed by 5 gram oral food challenges to walnut and the second tree nut (at 38 weeks). Unblinding to treatment group occurs at week 38, and active (walnut OIT) treatment subjects will continue on open-label walnut OIT maintenance dosing daily for up to a total of 298 weeks of therapy. Subjects reaching a qualifying specific IgE to walnut and the test tree nut at any early time point will receive a tolerance oral food challenge to the tree nuts on and 4 weeks off therapy. All subjects will have an oral food challenge on and off therapy at 142 weeks and at 298 weeks.
- Oat Powder: Oat Powder (placebo): Subjects randomized to the placebo (oat flour) group will undergo the same one-day desensitization protocol as the active (walnut) treatment group, consuming a maximum dose of 6 mg of oat powder (initial day escalation phase). After the initial escalation day achieving at least 1.5 mg and up to 6 mg of oat powder, the dosing build-up will occur every two weeks through dose 24 (1500mg oat flour) at ~34 weeks. A maintenance dose will be given for 4 weeks followed by a 5 gram protein OFC to walnut and a 5 gram protein OFC to a second tree nut (at ~38 weeks). Unblinding to treatment group occurs at week 38, and placebo subjects will be crossed over to active treatment with open-label walnut OIT with the same protocol as outlined for the active treatment group for up to 298 weeks of treatment beginning with initial escalation day.
Period: Overall Study
Arm/Group | Walnut Protein Powder | Oat Powder
Started | 10 | 4
Completed | 8 | 3
Not Completed | 2 | 1
Not completed — anxiety | 1 | 1
Not completed — diagnosis of ulcerative colitis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Walnut Protein Powder: 146 weeks for active treatment subjects
  Walnut Protein Powder: Dosing begins with a one-day walnut oral desensitization protocol. Starting at 0.1 mg protein and increasing every thirty minutes until a maximum dose of 6 mg is reached or until allergic symptoms develop. After the initial escalation day, subjects will continue daily dosing with dosing build-every two weeks to a maximum dose of 1500mg walnut protein at 34 weeks. A daily maintenance dose (1500mg or the highest dose reached by 34 weeks) will be given for 4 weeks followed by 5 gram oral food challenges to walnut and the second tree nut (at 38 weeks). Active treatment subjects will continue on maintenance dosing for up to a total of 298 weeks of therapy. Subjects reaching a qualifying specific IgE to walnut and the test tree nut at any early time point will receive a tolerance oral food challenge to the tree nuts on and 4 weeks off therapy. All subjects will have an oral food challenge on and off therapy at 142 weeks and at 298 weeks.
- Oat Powder: 184 weeks for placebo
  Oat Powder (placebo): Subjects in the placebo group will undergo the same one-day desensitization protocol as the active treatment group, consuming a maximum dose of 6 mg of oat powder (initial day escalation phase). After the initial escalation day achieving at least 1.5 mg and up to 6 mg of oat powder, the dosing build-up will occur every two weeks through dose 24 (1500mg oat flour) at ~34 weeks. A maintenance dose will be given for 4 weeks followed by a 5 gram protein OFC to walnut and a 5 gram protein OFC to a second tree nut (at ~38 weeks). Placebo subjects that fail the OFC will be crossed over to active treatment beginning with initial escalation day.
- Total: Total of all reporting groups
Arm/Group | Walnut Protein Powder | Oat Powder | Total
Number analyzed (Participants) | 10 | 4 | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8.7 [7.7 to 10] | 9.2 [8.9 to 9.8] | 9 [7 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 2 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 4 | 14
subjects with asthma [Number; unit: participants] | 3 | 3 | 6
subjects with atopic dermatitis [Number; unit: participants] | 6 | 4 | 10
subjects with allergic rhinitis [Number; unit: participants] | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Walnut OIT on Clinical Desensitization to Test Tree Nut as Measured by Change in Cumulative Tolerated Dose From Baseline to Week 38 at Oral Food Challenge
Description: Determine in tree nut allergic subjects the effectiveness of walnut oral immunotherapy on clinical desensitization to a second tree nut ("test tree nut") causing allergy when compared to placebo treatment, as measured by the change in cumulative dose from baseline oral food challenge (OFC) to the OFC to the test tree nut at approximately 38 weeks on therapy.
Time Frame: 38 weeks of therapy
Population: Participants completing the 38 week food challenge assessment were included in the analysis of primary outcome which was change in the cumulative tolerated dose during food challenge from baseline to week 38.
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Walnut Protein Powder | Oat Powder
Number analyzed (Participants) | 8 | 4
grams | 2.6 [1.55 to 3.54] | 0.05 [-0.47 to 0.17]
Statistical Analysis 1: Comparison: Walnut Protein Powder vs Oat Powder; Test type: Superiority — The change from baseline OFC to week 38 OFC (primary outcome measure) was compared between the two groups using a Mann-Whitney U test; p = 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Evaluation of Desensitization to Walnut Protein as Measured by Change in Cumulative Tolerated Dose From Baseline to Week 38 Oral Food Challenge
Description: Determine in tree nut allergic subjects the effectiveness of walnut oral immunotherapy on clinical desensitization to walnut causing allergy when compared to placebo treatment, as measured by the change in cumulative dose from baseline oral food challenge (OFC) to the OFC to the walnut at approximately 38 weeks on therapy.
Time Frame: 38 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Walnut Protein Powder | Oat Powder
Number analyzed (Participants) | 8 | 4
grams | 4.4 [3.1 to 4.9] | 0.6 [0.12 to 1.35]
Statistical Analysis 1: Comparison: Walnut Protein Powder vs Oat Powder; Test type: Superiority — Differences in dichotomous outcomes for the percentage of participants who reach the 5000 mg cumulative dose to the walnut at the week 38 desensitization OFC was analyzed using Fisher's exact test; p = 0.01, Fisher Exact

3. Secondary Outcome: Number (Percentage) of Subjects Reaching a Cumulative Tolerated Dose of 2000mg Walnut Protein at Desensitization OFC at Week 38
Description: The percentage of subjects reaching a cumulative protein dose of 2000mg at the desensitization oral food challenge to walnut at week 38
Time Frame: 38 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Oat Powder: Oat Powder (placebo): Subjects in the placebo group will undergo the same one-day desensitization protocol as the active treatment group, consuming a maximum dose of 6 mg of oat powder (initial day escalation phase). After the initial escalation day achieving at least 1.5 mg and up to 6 mg of oat powder, the dosing build-up will occur every two weeks through dose 24 (1500mg oat flour) at ~34 weeks. A maintenance dose will be given for 4 weeks followed by a 5 gram protein OFC to walnut and a 5 gram protein OFC to a second tree nut (at ~38 weeks). Placebo subjects that fail the OFC will be crossed over to active treatment beginning with initial escalation day.
Arm/Group | Walnut Protein Powder | Oat Powder
Number analyzed (Participants) | 8 | 4
Participants | 6 | 0
Statistical Analysis 1: Comparison: Walnut Protein Powder vs Oat Powder; Test type: Superiority — Differences in dichotomous outcomes including the percentage of subjects who reach the 2000 mg cumulative dose to the walnut at the week 38 desensitization OFC was analyzed using Fisher's exact test; p < 0.01, Fisher Exact

4. Secondary Outcome: Number (Percentage) of Subjects Reaching a Cumulative Tolerated Dose of 2000mg Test Tree Nut Protein at Desensitization OFC at Week 38
Description: Comparison of the number and percentage of subjects in each treatment arm reaching a cumulative protein dose of 2000mg at the week 38 (desensitization) oral food challenge to test tree nut
Time Frame: 38 weeks
Population: Participants completing the week 38 food challenge assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Walnut Protein Powder | Oat Powder
Number analyzed (Participants) | 8 | 4
Participants | 6 | 0
Statistical Analysis 1: Comparison: Walnut Protein Powder vs Oat Powder; Test type: Superiority — Differences in dichotomous outcomes such as the percentage of subjects who reach the 2000 mg cumulative dose to the tree nut at the week 38 desensitization OFC was analyzed using Fisher's exact test; p < 0.01, Fisher Exact

5. Secondary Outcome: Number (Percentage) of Subjects Attaining Sustained Unresponsiveness to Walnut and Test Tree Nut Proteins at Week 298 Oral Food Challenge
Description: The percentage of subjects demonstrating sustained unresponsiveness to walnut and to the test tree nut by end of study.
  Analysis group combines both active and placebo-crossover participants during open-label extension arm through the end of study at week 298. Subjects were able to exit the study at assessment timepoints earlier than week 298 if they are able to pass the sustained unresponsiveness oral food challenge, thus the analysis included all subjects through week 298..
Time Frame: up to 298 weeks on active treatment
Population: Those reaching sustained unresponsiveness to walnut and the test tree nut during open-label treatment by the end of study at week 298.
Measure: Count of Participants; unit: Participants
Groups:
- Open-label Walnut Protein Powder: up to 298 weeks of total active treatment
  Open-label treatment phase using walnut protein powder following unblinding of treatment arms after the 38 week oral food challenges. Active treatment subjects continued on open-label maintenance dosing for up to a total of 298 weeks of therapy. Placebo treatment subjects crossed over to active treatment following the active treatment protocol with 38 week oral food challenge assessment then continued open label maintenance dosing for upt to 298 weeks of therapy. Subjects reaching a qualifying specific IgE to walnut and the test tree nut at any early time point will receive a tolerance oral food challenge to the tree nuts on and 4 weeks off therapy. All subjects will have an oral food challenge on and off therapy at 142 weeks and at 298 weeks.
Arm/Group | Open-label Walnut Protein Powder
Number analyzed (Participants) | 11
Participants | 5

6. Secondary Outcome: Change in Skin Prick Test Wheal Size From Baseline to Week 142 in Active and Placebo Cross-over Subjects Receiving Active Walnut OIT
Description: Evaluation of walnut OIT on the mast cell responses as measured through change in skin prick testing to walnut in participants who were treated with walnut OIT to week 142. Analysis group combines both active and placebo-crossover participants from baseline through open-label treatment phase until the end of study.
Time Frame: 142 weeks
Population: Population analyzed combines active and placebo-crossover participants in the open-label phase of active walnut OIT. Change in skin test wheal size was measured from baseline to week 142 on active therapy. Baseline was defined for each arm as start of active treatment (active day=day 1; placebo arm (placebo cross-over)=week 38 (at start of active treatment period).
Measure: Median (Inter-Quartile Range); unit: mm wheal size
Groups:
- Open-label Walnut Protein Powder: Subjects tested at baseline and after 142 weeks of open-label WOIT for median skin prick test wheal size
Arm/Group | Open-label Walnut Protein Powder
Number analyzed (Participants) | 9
mm wheal size | 3.4 [0.8 to 4]
Statistical Analysis 1: Comparison: Open-label Walnut Protein Powder; Test type: Superiority; p < 0.001, Fisher Exact

7. Secondary Outcome: Serious Adverse Events Related to Walnut OIT Treatment
Description: Incidence of treatment-related serious adverse events during the study
Time Frame: 298 weeks active treatment
Population: All participants from study enrollment through blinded treatment phase at week 38, to open-label treatment through until exit of study, up to week 298.
Measure: Count of Participants; unit: Participants
Groups:
- Walnut Protein Powder: Walnut Protein Powder: Blinded study product dosing begins with a one-day walnut oral desensitization protocol. Starting at 0.1 mg protein and increasing every thirty minutes until a maximum dose of 6 mg is reached or until allergic symptoms develop. After the initial escalation day, subjects will continue daily dosing with dosing build-every two weeks to a maximum dose of 1500mg walnut protein at 34 weeks. A daily maintenance dose (1500mg or the highest dose reached by 34 weeks) will be given for 4 weeks followed by 5 gram oral food challenges to walnut and the second tree nut (at 38 weeks). Unblinding to treatment group occurs at week 38, and active treatment will continue on open-label daily maintenance dosing for up to a total of 298 weeks of therapy. Subjects reaching a qualifying specific IgE to walnut and the test tree nut at any early time point will receive a tolerance oral food challenge to the tree nuts on and 4 weeks off therapy. All subjects will have an oral food challenge on and off therapy at 142 weeks and at 298 weeks.
- Oat Powder: Oat Powder (placebo): Subjects randomized to the placebo group will undergo the same one-day desensitization protocol as the active treatment group, consuming a maximum dose of 6 mg of oat powder (initial day escalation phase). After the initial escalation day achieving at least 1.5 mg and up to 6 mg of oat powder, the dosing build-up will occur every two weeks through dose 24 (1500mg oat flour) at ~34 weeks. A maintenance dose will be given for 4 weeks followed by a 5 gram protein OFC to walnut and a 5 gram protein OFC to a second tree nut (at ~38 weeks). Placebo subjects will cross over to open-label active treatment at week 38 beginning with initial escalation day and following the same protocol as defined for active/walnut OIT for up to 298 weeks of active OIT.
- Open-label Walnut Protein Powder: This is the open-label phase of active dosing following the blinded treatment protocol through week 38. Following treatment unblinding at week 38, subjects on active treatment continued on daily maintenance treatment and those on placebo crossed over to active therapy per study protocol. All subjects in the open-label dosing phase were continued until the end of study at week 298 unless early exit criteria satisfied or the subject discontinued from the study.
Arm/Group | Walnut Protein Powder | Oat Powder | Open-label Walnut Protein Powder
Number analyzed (Participants) | 10 | 4 | 13
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first participant enrollment (April 2012) through last participant exit visit (May 2018). Maximum total engagement in the study for each participant was 298 weeks of active treatment (~6 years); however, study discontinuation could occur yearly depending on study outcome measures reached for each participant.
Description: SAE's are defined as per clinicaltrials.gov AE's included all events that were unrelated and related to OIT dosing with symptoms occurring within 2 hours of dosing or 2 hours after conclusion of study procedures (DPBCFC).
  Home OIT dose-related events, and treatment provided, were captured by daily, handwritten diary reporting by parents/participants AEs reported reflect entire trial with active and placebo-crossover subjects reported during blinded and open label stages
Groups:
- Walnut Protein Powder: 38 weeks for active treatment subjects
  Walnut Protein Powder: Blinded study product dosing begins with a one-day oral desensitization protocol. Starting at 0.1 mg protein and increasing every thirty minutes until a maximum dose of 6 mg is reached or until allergic symptoms develop. After the initial escalation day, subjects will continue daily dosing with dosing build-every two weeks to a maximum dose of 1500mg walnut protein at 34 weeks. A daily maintenance dose (1500mg or the highest dose reached by 34 weeks) will be given for 4 weeks followed by 5 gram oral food challenges to walnut and the second tree nut (at 38 weeks).
- Oat Powder: 38 weeks for placebo treatment subjects
  Oat Powder (placebo): Subjects in the placebo group will undergo the same one-day desensitization protocol as the active treatment group, consuming a maximum dose of 6 mg of oat powder (initial day escalation phase). After the initial escalation day achieving at least 1.5 mg and up to 6 mg of oat powder, the dosing build-up will occur every two weeks through dose 24 (1500mg oat flour) at ~34 weeks. A maintenance dose will be given for 4 weeks followed by a 5 gram protein OFC to walnut and a 5 gram protein OFC to a second tree nut (at ~38 weeks).
- Open-Label Walnut Protein Powder: Open-label treatment up to 298 weeks of active treatment
  Unblinding to treatment assignment occurs at week 38, and active treatment subjects continue on open-label, daily maintenance dosing for up to a total of 298 weeks of active therapy. Placebo subjects are crossed over to open-label, active treatment beginning using the dosing protocol for active treatment with OFC at week 38. Active treatment for all subjects is up to week 298. Subjects reaching a qualifying specific IgE to walnut and the test tree nut at any early time point will receive a tolerance oral food challenge to the tree nuts on and 4 weeks off therapy. All subjects will have an oral food challenge on and off therapy at 142 weeks and at 298 weeks.
Arm/Group | Walnut Protein Powder | Oat Powder | Open-Label Walnut Protein Powder
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/4 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/4 | 0/13
Other Adverse Events (participants affected / at risk) | 9/10 | 1/4 | 11/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Walnut Protein Powder (N=10) | Oat Powder (N=4) | Open-Label Walnut Protein Powder (N=13)
Concurrent illness/condition - not dose-related (Infections and infestations) | 3 (6) | 1 (3) | 11 (98)
Pre-existing disease or condition - not dose-related (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Concomitant medication - dose-related (Product Issues) | 0 (0) | 0 (0) | 0 (0) — Dose-related, AE-related epinephrine use
Abdominal pain - not dose-related (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
nasal congestion - dose-related (General disorders) | 4 (5) | 0 (0) | 1 (1)
flushing - dose related (Skin and subcutaneous tissue disorders) | 1 (13) | 1 (1) | 3 (7) — Symptoms related to OIT dose
cough - dose-related (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 0 (0) | 1 (1) — Symptoms related to OIT dose
abdominal pain - dose-related (Gastrointestinal disorders) | 7 (22) | 0 (0) | 6 (22)
throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — Symptoms related to OIT dose
rhinorrhea/sneezing - dose related (Respiratory, thoracic and mediastinal disorders) | 2 (7) | 0 (0) | 4 (6) — Symptoms related to OIT dose
mouth pruritus - dose-related (Gastrointestinal disorders) | 6 (17) | 0 (0) | 5 (11) — Symptoms related to OIT dose
Hives - dose-related (Skin and subcutaneous tissue disorders) | 3 (12) | 0 (0) | 2 (4) — Symptoms related to OIT dose
vomiting - dose-related (Gastrointestinal disorders) | 1 (4) | 0 (0) | 2 (3) — Symptoms related to OIT dose
Throat discomfort/pruritus (Respiratory, thoracic and mediastinal disorders) | 4 (50) | 0 (0) | 7 (14) — Symptoms related to dosing

LIMITATIONS AND CAVEATS:
Small sample size High screen failure rate High level of oropharyngeal symptoms Anxiety resulting in early termination Dosing fatigue with daily dosing Requirement for multiple food challenges in multi-tree nut assessment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes